CLINICAL TRIAL: NCT05938101
Title: Pain Clinic Staff Harassment Caused by Patients Pre/Post COVID Pandemic
Brief Title: Pain Clinic Staff Harassed by Patients Pre/Post COVID
Status: Recruiting | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: Salem2021 Harass PrePst COVID
Record Dates: First submitted 2023-07-06; First posted 2023-07-10 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Patient Violence
Keywords: Harassment by patient
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Behavioral therapy — Behavioral therapy and psychotherapy

SUMMARY:
Chronic pain may cause psychological or behavioral problems. Chronic pain patients occasionally harass the pain care providers. The COVID-19 pandemic caused major stress for the general population.

Quantitative and qualitative analysis of prospective electronic and clinic diary data. Evaluation of incidents of clinic staff harassment; caused by patients, before and during COVID pandemic. Analysis of causative factors, incident outcome and lessons learned.

DETAILED DESCRIPTION:
Chronic pain may be complicated by mental disease. Some patients have behavioral disorders and occasionally harass the pain care providers. The COVID-19 pandemic caused significant stress for the general population. The stress of the pandemic may aggravate the psychological dysfunction in chronic pain patients.

This is a quantitative and qualitative analysis of prospective electronic and clinic diary data. It is an evaluation of incidents of pain clinic staff harassment; caused by patients, before and during the COVID pandemic. This is an analysis of incident causative factors, incident outcomes, systemic factors and lessons learned. The qualitative information of each incident is presented in a sensitive and careful format.

ELIGIBILITY:
Inclusion Criteria:

* adult chronic pain patients

Exclusion Criteria:

* pediatric chronic pain patients

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult chronic pain patients who are undergoing treatment in a specialist pain clinic
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who harassed clinic staff | 12 months
  Percentage of patients who harassed clinic staff

CONTACTS AND LOCATIONS:
Overall Officials: Olu Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caruso R, Toffanin T, Folesani F, Biancosino B, Romagnolo F, Riba MB, McFarland D, Palagini L, Belvederi Murri M, Zerbinati L, Grassi L. Violence Against Physicians in the Workplace: Trends, Causes, Consequences, and Strategies for Intervention. Curr Psychiatry Rep. 2022 Dec;24(12):911-924. doi: 10.1007/s11920-022-01398-1. Epub 2022 Nov 29. PMID 36445636